CLINICAL TRIAL: NCT06737549
Title: Effect of Specific Mode Electroacupuncture Stimulation Combined with NGF on Dysphagia After Ischaemic Stroke: a Pilot Randomized Controlled Trial
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Xianming Lin, PHD, The Third Affiliated hospital of Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZSLL-KY-2024-074-01
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Ischemic Stroke; Dysphagia
MeSH Terms: conditions — Ischemic Stroke; Deglutition Disorders | interventions — Nerve Growth Factor; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- EA + NGF group (Experimental)
  Interventions: Drug: Nerver growth factor (NGF) injection; Device: EA intervention
- EA + placebo group (Placebo Comparator)
  Interventions: Drug: Placebo injection; Device: EA intervention
- Acupuncture + NGF group (Sham Comparator)
  Interventions: Drug: Nerver growth factor (NGF) injection; Device: Acupuncture intervention
- Acupuncture + placebo group (Sham Comparator)
  Interventions: Drug: Placebo injection; Device: Acupuncture intervention

INTERVENTIONS:
Drug: Nerver growth factor (NGF) injection — The 20ug mouse nerve growth factor (NO. S20060051, Jinlujie) will be obtained from Hiteck Biopharmaceutical Co., Ltd., Wuhan, China. mNGF will be dissolved in 2 ml of sterile water for injection and then injected intramuscularly into the gluteal muscle, three times a week for 6 weeks.
  Arms: Acupuncture + NGF group; EA + NGF group
Drug: Placebo injection — Patients will receive 2ml volume of physiological saline (PS) injected intramuscularly into the gluteal muscle, three times a week for 6 weeks.
  Arms: Acupuncture + placebo group; EA + placebo group
Device: EA intervention — Patients take supine position. After skin disinfection with 75% ethanol routine disinfection, the stainless needle (size 0.25mm×40mm, Hwato brand, Suzhou Medical Supplies Company Ltd in Jiangsu, China) will be inserted in GV20（Baihui) and the stainless needle(size 0.25mm×25mm, described above) will be inserted in GV26 (Shuigou), acupoints will be stimulated manually until patients feel soreness, distension or heaviness (the reaction of "De Qi"). Then, the needles are stimulated by using an acupuncture point nerve stimulator (HANS-200, Nanjing Jisheng, Ltd., China) with a frequency of 2/100 Hz and an intensity of patient can tolerate, targeting a current strength of 3.0mA, for 40 min (a homemade relay cycled power to the electrode for 6 sec on and 6 sec off), three times a week for 6 weeks.
  Arms: EA + NGF group; EA + placebo group
Device: Acupuncture intervention — Patients take supine position. After skin disinfection with 75% ethanol routine disinfection, the stainless needle (size 0.25mm×40mm, Hwato brand, Suzhou Medical Supplies Company Ltd in Jiangsu, China) will be inserted in GV20（Baihui) and the stainless needle(size 0.25mm×25mm, described above) will be inserted in GV26 (Shuigou), acupoints will be stimulated manually until patients feel soreness, distension or heaviness (the reaction of "De Qi"). Then, the needles are connected to an acupuncture point nerve stimulator (HANS-200, Nanjing Jisheng, Ltd., China) without closed circuit, with a frequency of 2/100 Hz and an intensity of 3 mA for 40 min (a homemade relay cycled power to the electrode for 6 sec on and 6 sec off), three times a week for 6 weeks.
  Arms: Acupuncture + NGF group; Acupuncture + placebo group

SUMMARY:
Ischemic stroke is a common clinical disease, often accompanied by dysphagia. At present, clinical treatment for patients with dysphagia after ischemic stroke is limited. The emergence of NGF has surprised the field of neurorehabilitation, but the clinical effect is not satisfactory. The main problem is that NGF is a macromolecular material with a molecular weight of 13.4 KD, which is difficult to penetrate the blood brain barrier. A large number of previous studies in our team have found that electroacupuncture with specific stimulation mode can open the blood brain barrier and induce NGF into the brain. Therefore, the purpose of this study is to investigate the effect of specific mode electroacupuncture stimulation combined with NGF treatment on patients with dysphagia after ischemic stroke and to explore the mechanism of this combination therapy to improve brain function, which creates a new method and theoretical basis for nerve rehabilitation of integrated traditional Chinese and Western medicine.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with first-ever ischemic stroke confirmed by Computed Tomography (CT) and/or Magnetic Resonance Imaging (MRI);
2. Onset time ranged from 15 days to 180 days;
3. Aged 18 to 80 years old, male or female;
4. Dysphagia confirmed by a videofluoroscopic swallowing study (VFSS);
5. Patients who are able to accept and comply with acupuncture, electroacupuncture treatment, gluteal intramuscular injection, and have good compliance;
6. Have provided signed consent and exhibit willingness to participate in the trial.
7. Women who are lactating, pregnant or intending to get pregnant;

Exclusion Criteria:

1. Patients with dysphagia before ischemic stroke onset or dysphagia not caused by ischemic stroke;
2. Patients with severe cognitive impairment;
3. Patients with severe cardiac, hepatic, and renal dysfunction, as well as severe coagulation abnormalities;
4. Patients with other abnormal test results who are deemed unsuitable to participate in this study by the investigator.
5. Multiple occurrences of stroke, or a history of craniocerebral surgery, or cerebral infarction caused by trauma or brain tumors.
6. Patients with severe neurological deficits prior to ischemic stroke, such as visual and auditory impairments, aphasia, agnosia, severe hemiplegia, and other conditions.
7. Women who are lactating, pregnant or intending to get pregnant;
8. Patients with a history of needle fainting or with skin infections at the acupuncture site.
9. Cardiac pacemaker carrier;
10. Patients allergic to NGF;
11. The inability to undergo VFSS;
12. Patients with a medication history that may alter cortical excitability within the past 2 months.
13. Patients who are currently participating in other clinical trials or have participated in clinical trials that ended within the last 3 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Functional Oral Intake Scale (FOIS) | week 0, week 2, week 4, week 6, week 12

SECONDARY OUTCOMES:
Dysphagia Outcome and Severity Scale (DOSS) | week 0, week 6
Penetration Aspiration Scale (PAS) | week 0, week 6
modified Rankin Scale (mRS) | week 0, week 2, week 4, week 6
Modified Barthel Index (MBI) | week 0, week 2, week 4, week 6
Oxygenated hemoglobin and deoxygenated hemoglobin in cerebral cortex | week 0, week 6
  Measure method: fNIRS

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
The data and results of this study need to be confirmed by Xianming Lin.

REFERENCES:
- [Background] Fu X, Li H, Yang W, Li X, Lu L, Guo H, Guo K, Huang Z. Electroacupuncture at HT5 + GB20 promotes brain remodeling and significantly improves swallowing function in patients with stroke. Front Neurosci. 2023 Nov 2;17:1274419. doi: 10.3389/fnins.2023.1274419. eCollection 2023. PMID 38027487
- [Background] Dai M, Qian K, Ye Q, Yang J, Gan L, Jia Z, Pan Z, Cai Q, Jiang T, Ma C, Lin X. Specific Mode Electroacupuncture Stimulation Mediates the Delivery of NGF Across the Hippocampus Blood-Brain Barrier Through p65-VEGFA-TJs to Improve the Cognitive Function of MCAO/R Convalescent Rats. Mol Neurobiol. 2025 Feb;62(2):1451-1466. doi: 10.1007/s12035-024-04337-8. Epub 2024 Jul 12. PMID 38995444
- [Background] Lin Y, Gan L, Ren L, Ma C, Dai M, Qian K, Ye Q, Lin X. Acupuncture with specific mode electro-stimulation effectively and transiently opens the BBB through Shh signaling pathway. Neuroreport. 2023 Dec 13;34(18):873-886. doi: 10.1097/WNR.0000000000001970. Epub 2023 Nov 8. PMID 37942738
- [Background] Sheng L, Yin L, Peng D, Zhao L. From Best Evidence to Best Practice: Enteral Nutrition from Continuous Nasal Feeding in Stroke Patients. Int J Gen Med. 2020 Oct 22;13:927-936. doi: 10.2147/IJGM.S269393. eCollection 2020. PMID 33132703
- [Background] Zhang H, Park JH, Maharjan S, Park JA, Choi KS, Park H, Jeong Y, Ahn JH, Kim IH, Lee JC, Cho JH, Lee IK, Lee CH, Hwang IK, Kim YM, Suh YG, Won MH, Kwon YG. Sac-1004, a vascular leakage blocker, reduces cerebral ischemia-reperfusion injury by suppressing blood-brain barrier disruption and inflammation. J Neuroinflammation. 2017 Jun 23;14(1):122. doi: 10.1186/s12974-017-0897-3. PMID 28645333
- [Background] Gutierrez-Fernandez M, Fuentes B, Rodriguez-Frutos B, Ramos-Cejudo J, Vallejo-Cremades MT, Diez-Tejedor E. Trophic factors and cell therapy to stimulate brain repair after ischaemic stroke. J Cell Mol Med. 2012 Oct;16(10):2280-90. doi: 10.1111/j.1582-4934.2012.01575.x. PMID 22452968
- [Background] Barbero P, Busso M, Tinivella M, Artusi CA, De Mercanti S, Cucci A, Veltri A, Avagnina P, Calvo A, Chio' A, Durelli L, Clerico M. Long-term follow-up of ultrasound-guided botulinum toxin-A injections for sialorrhea in neurological dysphagia. J Neurol. 2015 Dec;262(12):2662-7. doi: 10.1007/s00415-015-7894-1. Epub 2015 Sep 26. PMID 26410746
- [Background] Rofes L, Muriana D, Palomeras E, Vilardell N, Palomera E, Alvarez-Berdugo D, Casado V, Clave P. Prevalence, risk factors and complications of oropharyngeal dysphagia in stroke patients: A cohort study. Neurogastroenterol Motil. 2018 Mar 23:e13338. doi: 10.1111/nmo.13338. Online ahead of print. PMID 29573064
- [Background] Labeit B, Michou E, Hamdy S, Trapl-Grundschober M, Suntrup-Krueger S, Muhle P, Bath PM, Dziewas R. The assessment of dysphagia after stroke: state of the art and future directions. Lancet Neurol. 2023 Sep;22(9):858-870. doi: 10.1016/S1474-4422(23)00153-9. PMID 37596008